CLINICAL TRIAL: NCT00869674
Title: 一项比较GeneSearch 乳腺淋巴结（BLN）检测试剂盒和永久病理切片检测乳腺癌患者腋窝前哨淋巴结转移的前瞻性、多中心临床试验 A Prospective and Multi-center Clinical Trial By Comparing GeneSearch™ Breast Lymph Node (BLN) Test Kit To Permanent Pathological Section On Detecting Axillary Sentinel Lymph Node Metastases In Breast Cancer Patients
Brief Title: GeneSearch™ Breast Lymph Node (BLN) Assay China Registration Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Investigational products has been suspended from the US market
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OCD-200804; CBCSG-001a
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: GeneSearch; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biological Assay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine pathologic method (No Intervention): Half of each sentinal lymph node will have rountine pathologic examination as normal practice.
- GeneSearch BLN Assay (Experimental): Half of each sentinal lymph node will have GeneSearch BLN testing.
  Interventions: Procedure: GeneSearch™ Breast Lymph Node (BLN) Assay

INTERVENTIONS:
Procedure: GeneSearch™ Breast Lymph Node (BLN) Assay — Each of the sentinal lymph node will be divided in half according to cutting scheme.
  Half of the sentinal lymph node will be tested using rountine pathological method as normal practice, half of the node will have GeneSearch BLN testing.
  Other Names: GeneSearch; Pathology
  Arms: GeneSearch BLN Assay

SUMMARY:
The primary objective of this trial is to compare GeneSearch™ Breast Lymph Node (BLN) Test Kit to permanent pathological section, so as to evaluate the clinical sensitivity and specificity of GeneSearch™ Breast Lymph Node (BLN) Test Kit in detecting axillary sentinel lymph node metastases in breast cancer patients.

The secondary objective of this trial is to evaluate the positive predictive value and negative predictive value of GeneSearch™ Breast Lymph Node (BLN) Test Kit when used in the detection of axillary sentinel lymph node metastases in breast cancer patients.

Prospective and multi-center clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed previously as breast cancer
* patient scheduled for sentinel lymph node dissection
* 18 years or older
* female or male, and
* able and willing to give consent to participate in the study

Exclusion Criteria:

* Patients taking part in other research studies that would interfere with their full participation in this study, or
* Prior sentinel or partial axillary lymphadenectomy on the same body side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To compare GeneSearch™ BLN Test Kit to permanent pathological section to evaluate the clinical sensitivity and specificity of GeneSearch™ BLN Test Kit in detecting axillary sentinel lymph node metastases in breast cancer patients. | 9 months

SECONDARY OUTCOMES:
To evaluate the positive predictive value and negative predictive value of GeneSearch™ BLN Test Kit when used in the detection of axillary sentinel lymph node metastases in breast cancer patients. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangdong, Guangdong
  - Second affiliated hospital of Zhongshan University, Guangzhou, Guangdong
  - China Shandong Cancer hospital, Jinan, Shandong
  - Southwest Hospital, Chongqing, Sichuan
  - Shanghai Cancer Hospital, Shanghai

REFERENCES:
- [Background] Valagussa P, Bonadonna G, Veronesi U. Patterns of relapse and survival following radical mastectomy. Analysis of 716 consecutive patients. Cancer. 1978 Mar;41(3):1170-8. doi: 10.1002/1097-0142(197803)41:33.0.co;2-i. PMID 638961
- [Background] Fisher B, Bauer M, Wickerham DL, Redmond CK, Fisher ER, Cruz AB, Foster R, Gardner B, Lerner H, Margolese R, et al. Relation of number of positive axillary nodes to the prognosis of patients with primary breast cancer. An NSABP update. Cancer. 1983 Nov 1;52(9):1551-7. doi: 10.1002/1097-0142(19831101)52:93.0.co;2-3. PMID 6352003
- [Background] Albertini JJ, Lyman GH, Cox C, Yeatman T, Balducci L, Ku N, Shivers S, Berman C, Wells K, Rapaport D, Shons A, Horton J, Greenberg H, Nicosia S, Clark R, Cantor A, Reintgen DS. Lymphatic mapping and sentinel node biopsy in the patient with breast cancer. JAMA. 1996 Dec 11;276(22):1818-22. PMID 8946902
- [Background] Giuliano AE, Dale PS, Turner RR, Morton DL, Evans SW, Krasne DL. Improved axillary staging of breast cancer with sentinel lymphadenectomy. Ann Surg. 1995 Sep;222(3):394-9; discussion 399-401. doi: 10.1097/00000658-199509000-00016. PMID 7677468
- [Background] Morton DL. Intraoperative lymphatic mapping and sentinel lymphadenectomy: community standard care or clinical investigation? Cancer J Sci Am. 1997 Nov-Dec;3(6):328-30. No abstract available. PMID 9403042
- [Background] Yared MA, Middleton LP, Smith TL, Kim HW, Ross MI, Hunt KK, Sahin AA. Recommendations for sentinel lymph node processing in breast cancer. Am J Surg Pathol. 2002 Mar;26(3):377-82. doi: 10.1097/00000478-200203000-00013. PMID 11859211
- [Background] Schrenk P, Rieger R, Shamiyeh A, Wayand W. Morbidity following sentinel lymph node biopsy versus axillary lymph node dissection for patients with breast carcinoma. Cancer. 2000 Feb 1;88(3):608-14. doi: 10.1002/(sici)1097-0142(20000201)88:33.0.co;2-k. PMID 10649254
- [Background] Treseler PA, Tauchi PS. Pathologic analysis of the sentinel lymph node. Surg Clin North Am. 2000 Dec;80(6):1695-719. doi: 10.1016/s0039-6109(05)70256-5. PMID 11140868
- [Background] Van Diest PJ, Torrenga H, Borgstein PJ, Pijpers R, Bleichrodt RP, Rahusen FD, Meijer S. Reliability of intraoperative frozen section and imprint cytological investigation of sentinel lymph nodes in breast cancer. Histopathology. 1999 Jul;35(1):14-8. doi: 10.1046/j.1365-2559.1999.00667.x. PMID 10383709
- [Background] Veronesi U, Paganelli G, Galimberti V, Viale G, Zurrida S, Bedoni M, Costa A, de Cicco C, Geraghty JG, Luini A, Sacchini V, Veronesi P. Sentinel-node biopsy to avoid axillary dissection in breast cancer with clinically negative lymph-nodes. Lancet. 1997 Jun 28;349(9069):1864-7. doi: 10.1016/S0140-6736(97)01004-0. PMID 9217757
- [Background] Veronesi U, Paganelli G, Viale G, Galimberti V, Luini A, Zurrida S, Robertson C, Sacchini V, Veronesi P, Orvieto E, De Cicco C, Intra M, Tosi G, Scarpa D. Sentinel lymph node biopsy and axillary dissection in breast cancer: results in a large series. J Natl Cancer Inst. 1999 Feb 17;91(4):368-73. doi: 10.1093/jnci/91.4.368. PMID 10050871
- [Background] Viale G, Bosari S, Mazzarol G, Galimberti V, Luini A, Veronesi P, Paganelli G, Bedoni M, Orvieto E. Intraoperative examination of axillary sentinel lymph nodes in breast carcinoma patients. Cancer. 1999 Jun 1;85(11):2433-8. PMID 10357414
- [Background] Anderson TJ. The challenge of sentinel lymph node biopsy. Histopathology. 1999 Jul;35(1):82-4. doi: 10.1046/j.1365-2559.1999.00737.x. No abstract available. PMID 10383718
- [Background] Krag D. Current status of sentinel lymph node surgery for breast cancer. J Natl Cancer Inst. 1999 Feb 17;91(4):302-3. doi: 10.1093/jnci/91.4.302. No abstract available. PMID 10050858
- [Background] Turner RR, Hansen NM, Stern SL, Giuliano AE. Intraoperative examination of the sentinel lymph node for breast carcinoma staging. Am J Clin Pathol. 1999 Nov;112(5):627-34. doi: 10.1093/ajcp/112.5.627. PMID 10549249
- [Background] Lockett MA, Metcalf JS, Baron PL, O'Brien PH, Elliott BM, Robison JG, Cole DJ. Efficacy of reverse transcriptase-polymerase chain reaction screening for micrometastic disease in axillary lymph nodes of breast cancer patients. Am Surg. 1998 Jun;64(6):539-43; discussion 543-4. PMID 9619175
- [Background] Julian TB, Blumencranz P, Deck K, Whitworth P, Berry DA, Berry SM, Rosenberg A, Chagpar AB, Reintgen D, Beitsch P, Simmons R, Saha S, Mamounas EP, Giuliano A. Novel intraoperative molecular test for sentinel lymph node metastases in patients with early-stage breast cancer. J Clin Oncol. 2008 Jul 10;26(20):3338-45. doi: 10.1200/JCO.2007.14.0665. PMID 18612150
- [Background] Bernstein JL, Godbold JH, Raptis G, Watson MA, Levinson B, Aaronson SA, Fleming TP. Identification of mammaglobin as a novel serum marker for breast cancer. Clin Cancer Res. 2005 Sep 15;11(18):6528-35. doi: 10.1158/1078-0432.CCR-05-0415. PMID 16166429
- [Background] Zehentner BK, Carter D. Mammaglobin: a candidate diagnostic marker for breast cancer. Clin Biochem. 2004 Apr;37(4):249-57. doi: 10.1016/j.clinbiochem.2003.11.005. PMID 15003725
- [Background] Schoenfeld A, Kruger KH, Gomm J, Sinnett HD, Gazet JC, Sacks N, Bender HG, Luqmani Y, Coombes RC. The detection of micrometastases in the peripheral blood and bone marrow of patients with breast cancer using immunohistochemistry and reverse transcriptase polymerase chain reaction for keratin 19. Eur J Cancer. 1997 May;33(6):854-61. doi: 10.1016/s0959-8049(97)00014-2. PMID 9291805
- [Background] Backus J, Green GA, XU M, et al. Intra-operative molecular analysis of sentinel lymph nodes for the management of breast Cancer surgery. Clin Cancer Res; 2005
- [Background] Turner RR, Weaver DL, Cserni G, Lester SC, Hirsch K, Elashoff DA, Fitzgibbons PL, Viale G, Mazzarol G, Ibarra JA, Schnitt SJ, Giuliano AE. Nodal stage classification for breast carcinoma: improving interobserver reproducibility through standardized histologic criteria and image-based training. J Clin Oncol. 2008 Jan 10;26(2):258-63. doi: 10.1200/JCO.2007.13.0179. PMID 18182666
- [Derived] Liu YH, Xu FP, Liao N, Li L, Zhang GC, Zhuang HG, Mei P, Xu J, Zhu XL, Luo XL, Kuang LJ. Efficacy of intraoperative GeneSearch Breast Lymph Node (BLN) Assay for breast cancer metastasis detection in sentinel lymph node in Chinese patients. Cancer Sci. 2010 Aug;101(8):1920-4. doi: 10.1111/j.1349-7006.2010.01618.x. Epub 2010 Jan 17. PMID 20557308